CLINICAL TRIAL: NCT06300073
Title: Plaque Removal Efficacy of AutoBrush®, a 360 Degree Sonic Power Toothbrush in Children
Brief Title: Plaque Removal Efficacy of a U-Shaped Sonic Power Toothbrush in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lander Enterprises, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AB-360-001-2022
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Dental Plaque
Keywords: gingivitis; toothbrush
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: single-use, randomized, two-period, cross-over study
Who Masked: Outcomes Assessor
Masking Description: Examiner and data recorder will not have access to the room for test materials dispensing and instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AutoBrush U-shaped power toothbrush, then Manual Toothbrush (Experimental): Participants first received the AutoBrush U-shaped power toothbrush with fluoride toothpaste for a single brushing use for 30 seconds; after a 2-day washout period, participants received the ADA reference manual toothbrush for a single brushing use for 2 minutes.
  Interventions: Device: Experimental: U-shaped Power Toothbrush; Device: Placebo Comparator: Soft Manual Toothbrush
- Manual Toothbrush (Experimental): Participants first received the ADA reference manual toothbrush for a single brushing use for 2 minutes; after a 2-day washout period, participants received the AutoBrush U-shaped power toothbrush with fluoride toothpaste for a single brushing use for 30 seconds.
  Interventions: Device: Experimental: U-shaped Power Toothbrush; Device: Placebo Comparator: Soft Manual Toothbrush

INTERVENTIONS:
Device: Experimental: U-shaped Power Toothbrush — Twice daily brushing for 30 seconds with fluoride toothpaste
Device: Placebo Comparator: Soft Manual Toothbrush — Twice daily brushing for 2 minutes with fluoride toothpaste

SUMMARY:
The objective of this single-use, examiner blinded, randomized, two-period, cross-over, IRB-approved clinical study is to evaluate the safety and plaque removal efficacy of AutoBrush®, a new children's 360° sonic toothbrush, compared to a marketed children's manual toothbrush.

DETAILED DESCRIPTION:
Up to 22 healthy children (5-8 years old) will be enrolled in a single-center, single-use, randomized, two-period, IRB approved cross-over study. Subjects will be randomly assigned to one of two treatment sequences: 1) brush two minutes with marketed children's manual toothbrush (MTB) or 2) brush 30 seconds with AutoBrush® 360° Sonic Toothbrush (AB) and fluoride toothpaste. Qualified subjects will have pre-brushing supragingival plaque levels ≥ 1.8 according to the Lobene-Soparkar Modified Turesky Modification of the Quigley-Hein Plaque Index (PI), following 12-16 hours plaque accumulation period. Under parent's supervision, subjects brushed at home with their assigned toothbrush, twice daily during a 2-day familiarization period. After refraining (12-16 hours) from oral hygiene, subjects returned for plaque assessment, supervised use of their assigned toothbrush and a post-brushing plaque evaluation. Subjects were given the second toothbrush to begin the next 2-day familiarization period and second period evaluation procedures. Analysis of covariance (ANCOVA) will be used for single-use brushing PI models to assess whole mouth and 8 other hard-to-reach tooth sites.

ELIGIBILITY:
To be eligible for study participation, subjects must meet the following criteria:

1. Generally healthy males and females at least 5-8 years of age.
2. Volunteers provide assent to participate and consent from a parent or legal guardian prior to being enrolled into the study.
3. A minimum of 12 natural teeth with scorable facial and lingual surfaces. Partially erupted permanent teeth and primary teeth that are loose or in the process of exfoliation are not included in the tooth count. Teeth that ware grossly carious, orthodontically banded, exhibiting general cervical abrasion and/or enamel abrasion ware not included in the tooth count.
4. A plaque index score ≥ 1.80 according to the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index, following 12 to 16 hours plaque accumulation

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Having a history of adverse effects, oral soft or hard tissue sensitivity, to any ingredient in the test materials.
2. Having self-reported serious medical conditions.
3. Being under treatment for a heart condition requiring use of a pacemaker.
4. Having anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
5. Having had antibiotic, anti-inflammatory, anti-coagulant medication or chemotherapeutic antiplaque/antigingivitis therapy within 30 days of screening exams.
6. Having participated in any study involving oral care products, concurrently or within the 30 days of screening exams.
7. Presence of severe periodontal disease or being actively treated for periodontal disease.
8. Having grossly carious, fully crowned, or extensively restored teeth.
9. Having orthodontic appliances, peri/oral piercings, or removable partial dentures.
10. Having significant oral soft tissue pathology based on a visual examination.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Within-Treatment Whole-Mouth Differences (vs Baseline) - Plaque removal Mean Change from baseline (pre-brushing to post-brushing) in plaque score after single supervised use based on all tooth surfaces of the whole mouth. | Up to 2 weeks
  Supragingival dental plaque: Lobene-Soparkar Modification of Turesky Modification of Quigley-Hein Plaque Index
  Plaque will be disclosed using a red disclosing solution and each tooth will be scored in six areas (disto-buccal, mid-buccal and mesio-buccal, disto-lingual, mid-lingual and mesio-lingual), according to the criteria noted below:
  0 = No plaque.
  1. = Separate flecks or discontinuous band of plaque at the gingival (cervical) margin.
  2. = Thin (up to 1 mm), continuous band of plaque at the gingival margin.
  3. = Band of plaque wider than 1 mm but less than 1/3 of tooth surface area.
  4. = Plaque covering 1/3 or more, but less than 2/3 of tooth surface area.
  5. = Plaque covering 2/3 or more of tooth surface area.

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Inc, Fort Wayne, Indiana, United States